CLINICAL TRIAL: NCT03018847
Title: Evaluation of COPD Co-Pilot
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: HGE Health Care Solutions, LLC (Industry)
Collaborators: PneumRx, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CPV2-2016-S1
Record Dates: First submitted 2017-01-10; First posted 2017-01-12 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: COPD Co-Pilot — The COPD Co-Pilot is a system that guides a patient through a software application (web or mobile app) to collect, track, and trend daily symptoms related to Chronic Obstructive Pulmonary Disease (COPD). The system is intended to be used by patients as a support tool to track COPD symptoms as part of their personal disease management plan. The COPD Co-Pilot allows health care providers to view and triage subject symptoms via the provider web-based application. Health care providers also have the ability to send responses to subjects, like medication recommendations, through preset forms in the system.

SUMMARY:
The purpose of undertaking this study is to examine the use of COPD Co-PilotTM, a COPD disease management program manufactured and operated by HGE Health Care Solutions, LLC, in COPD patients outside of the geographic base of HGE's existing patient population (Philadelphia, PA). The purpose is to demonstrate the feasibility of expanding the program to additional geographic sites and to examine whether similar outcome measures are achieved in patients under the supervision of health care providers that are new to the program.

.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has read, understood and signed an informed consent form prior to enrollment.
2. Males or females age ≥35 years old
3. Documented diagnosis of moderate to very severe COPD (GOLD Level II-IV)
4. Must be able to read and understand English and consent for themselves
5. Subject is willing and able to use an iPad mini device.

Exclusion Criteria:

1. Subject has a cognitive impairment (determined by physician) that will make it hard to follow instructions regarding device usage
2. Subject is currently known to suffer from or have a history of significant substance abuse within the last 2 years
3. Subject has any condition that in the opinion of the provider may adversely affect their participation
4. Subject is residing in hospice care, Skilled Nursing Facilities or Long Term Acute Care facilities
5. Subject has a planned procedures at time of enrollment that will occur within timeframe of study that will require hospitalization or otherwise adversely affect their ability to participate
6. Subject has no cellular coverage at their primary residence
7. Subject plans to travel to a location with no cellular coverage for a significant period (>1 week) during their program participation

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects shall be recruited from the pool of patients at the investigative site that have been diagnosed with moderate to severe COPD.
  The study is planned to enroll 100 subjects. The study will be conducted at one investigative site in the United States, the Medical University of South Carolina Health System. Recruitment will stop when 100 subjects are enrolled. There will be no replacement for dropouts. Recruitment is planned to last approximately 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2017-01; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Patient Adoption | 6 months
  Percentage of potential daily symptom reports completed by patients

SECONDARY OUTCOMES:
Patient Satisfaction | 6 months
  patient satisfaction questionnaire
Inpatient Admissions | 6 months
  admission records for period prior to study and during study
Emergency department visits | 6 months
  emergency department records for period prior to study and during study
Clinic visits | 6 months
  clinic visits for period prior to study and during study
Patient reported respiratory symptoms | 6 months
  Daily values for breathlessness, sputum quantity, sputum color, sputum consistency, peak flow, temperature over 100 F, cough, wheeze, sore throat, and nasal congestion.
Symptom change detected | 6 months
  Change index (a numeric value) and the categorical level of change that corresponds to the patient's reported symptoms when compared to their baseline. This is recorded for each daily symptom report submitted after completion of the run-in period.
Episode duration | 6 months
  the date when a mild, moderate or significant level of change is first detected for a patient through the date immediately followed by seven consecutive days in which no level of change is detected. The total number of days in this period, symptoms reported during this period, and clinical responses communicated to the patient (including any treatments or changes) will be reported for analysis.
Clinical responses | 6 months
  the date, medication or instruction, dosage, frequency, duration of clinical responses sent to subjects, and time elapsed between the patient's check-in and the time the response was acknowledged by the patient.
Hospitalization history | 6 months
  hospitalization history reported to Health Assistants by patients during scheduled monthly phone calls. This will be reconciled with admissions data from the site and may include utilization at other institutions.
Medications | 6 months
  list of medications entered by site coordinator, provider, or reported by subjects to Health Assistants during scheduled monthly phone calls.
Patient profile information | 6 months
  This will include, among other variables, medial history, smoking history, spirometry results, oxygen use, and diagnoses of co-morbidities.
Medication compliance | 6 months
  compliance with newly prescribed treatments as reported by patients during follow up phone calls.
Length of stay | 6 months
  total number of inpatient days and the average length of stay per admission will be reported for analyses. These records will include date of admission, date of discharge, patient name and medical record number, patient date of birth (DOB), location, length of stay, attending physician, admission diagnosis and diagnosis at discharge. Reported for period prior to study and during study period
Readmissions | 6 months
  The number of inpatient admissions that occurred within 30, 60, and 90 days of discharge from a prior admission will be reported for analyses. These records will include date of admission, date of discharge, patient name and medical record number, patient DOB, location, length of stay, attending physician, admission diagnosis, diagnosis at discharge, and associated costs broken down by category. This will be reported for time prior to study and during study period.
Readmission rate | 6 months
  The rate and percent of inpatient admissions that occurred within 30, 60, and 90 days of discharge from a prior admission will be reported for analyses. These records will include date of admission, date of discharge, patient name and medical record number, patient DOB, location, length of stay, attending physician, admission diagnosis and diagnosis at discharge. These will be reported for the period prior to the start of the study through the study period.
Source of inpatient admissions and visits to the Emergency Department (ED) | 6 months
  The source (e.g. from home, from accident, from outpatient clinical, at direction of physician, from ED, etc.) of each and every inpatient admission an emergency department visit will be reported for analyses. These will be reported for the period prior to the enrollment through the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Tatsiana Beiko, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith HS, Criner AJ, Fehrle D, Grabianowski CL, Jacobs MR, Criner GJ. Use of a SmartPhone/Tablet-Based Bidirectional Telemedicine Disease Management Program Facilitates Early Detection and Treatment of COPD Exacerbation Symptoms. Telemed J E Health. 2016 May;22(5):395-9. doi: 10.1089/tmj.2015.0135. Epub 2015 Oct 9. PMID 26451903
- [Background] Cordova FC, Ciccolella D, Grabianowski C, Gaughan J, Brennan K, Goldstein F, Jacobs MR, Criner GJ. A Telemedicine-Based Intervention Reduces the Frequency and Severity of COPD Exacerbation Symptoms: A Randomized, Controlled Trial. Telemed J E Health. 2016 Feb;22(2):114-122. doi: 10.1089/tmj.2015.0035. Epub 2015 Aug 10. PMID 26259074
- [Background] Kim V, Garfield JL, Grabianowski CL, Krahnke JS, Gaughan JP, Jacobs MR, Criner GJ. The effect of chronic sputum production on respiratory symptoms in severe COPD. COPD. 2011 Apr;8(2):114-20. doi: 10.3109/15412555.2011.558546. PMID 21495839
- [Background] So JY, Lastra AC, Zhao H, Marchetti N, Criner GJ. Daily Peak Expiratory Flow Rate and Disease Instability in Chronic Obstructive Pulmonary Disease. Chronic Obstr Pulm Dis. 2015 Nov 11;3(1):398-405. doi: 10.15326/jcopdf.3.1.2015.0142. PMID 28848862
- [Background] Remakus, Christopher B., et al.